CLINICAL TRIAL: NCT05235581
Title: Study of the Postural Reactions of Balance Compared Between Real Environment and Virtual Environment With Avatar and Reinforced Visual Signal.
Brief Title: Balance Reactions in a Virtual Environment With Avatar and/or Reinforced Visual Signal Compared to a Real Environment
Acronym: EQUIVIRT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pôle Saint Hélier (Other)
Collaborators: Hopital La Musse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 2021-A01623-38
Record Dates: First submitted 2022-01-28; First posted 2022-02-11 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, controlled, randomized study on healthy volunteers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BCAD's arm (Experimental): The 4 interventions are in the BCAD's order.
  Interventions: Other: Intervention A : virtual environment with avatar; Other: Intervention B : virtual environment with reinforced visual signal; Other: Intervention C : virtual environment with avatar and reinforced visual signal; Other: Intervention D : real environment
- BACD's arm (Experimental): The 4 interventions are in the BACD's order.
  Interventions: Other: Intervention A : virtual environment with avatar; Other: Intervention B : virtual environment with reinforced visual signal; Other: Intervention C : virtual environment with avatar and reinforced visual signal; Other: Intervention D : real environment
- CABD's arm (Experimental): The 4 interventions are in the CABD's order.
  Interventions: Other: Intervention A : virtual environment with avatar; Other: Intervention B : virtual environment with reinforced visual signal; Other: Intervention C : virtual environment with avatar and reinforced visual signal; Other: Intervention D : real environment
- ACBD's arm (Experimental): The 4 interventions are in the ACBD's order.
  Interventions: Other: Intervention A : virtual environment with avatar; Other: Intervention B : virtual environment with reinforced visual signal; Other: Intervention C : virtual environment with avatar and reinforced visual signal; Other: Intervention D : real environment

INTERVENTIONS:
Other: Intervention A : virtual environment with avatar — 30-second right and left unipodal static and dynamic balance test with avatar only
Other: Intervention B : virtual environment with reinforced visual signal — 30-second right and left unipodal static and dynamic balance test with reinforced visual signal only
Other: Intervention C : virtual environment with avatar and reinforced visual signal — 30-second right and left unipodal static and dynamic balance test with avatar and reinforced visual signal
Other: Intervention D : real environment — 30-second right and left unipodal static and dynamic balance test in real environment

SUMMARY:
The scientific literature shows that there is a degradation of balance in virtual reality. This trial investigates the introduction of a full-body avatar and/or enhanced visual cues on the reduction of the degradation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer, men and women over 18 years old

Exclusion Criteria:

* Severe visual deficiency not allowing an activity in immersive virtual reality.
* Immobilization of one of the upper limbs (splint restraint splint)
* Orthopedic and painful problems of the inferior limb
* MSSQ greater than 25
* Pregnant woman
* Person under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
Area of CoP (Center of pression) for each test (in cm²) | Immediately after inclusion
  Mesure of area of center of pression during the balance tests in virtual condition and real condition, order in terms of randomisation
Total distance covered by the CoP during the balance test (in cm) | Immediately after inclusion
  Mesure of the total distance covered by the CoP during the balance tests (in cm) in virtual condition and real condition, order in terms of randomisation

SECONDARY OUTCOMES:
Simulator Sickness Quantifying (SSQ) | Immediately after the balance test
  SSQ completed after the balance test, SSQ is a scale of cyber sickness, from 0 to 48

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Pôle Saint Hélier, Rennes, Brittany Region
  - Hôpital la Musse, Saint-Sébastien-de-Morsent